CLINICAL TRIAL: NCT00762593
Title: A Multicenter Double Blind Randomized Placebo Controlled Trial Evaluating Transvaginal Electrical Stimulation With a Home Use Programmable Device for Urinary Stress Incontinence
Brief Title: Trial Evaluating Transvaginal Electrical Stimulation With a Home Use Programmable Device for Urinary Stress Incontinence
Acronym: KEAT F1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Akontis (Industry)
Responsible Party: Jacques Croissandeau, Akontis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KEAT F1
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Urinary Stress Incontinence
Keywords: urinary stress incontinence; urinary stress incontinence in women
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): transvaginal electrical stimulation with a home use programmable device used 30 minutes every day during 8 weeks
  Interventions: Device: transvaginal electrical stimulation device
- 2 (Placebo Comparator): Use of a transvaginal placebo home use programmable device used 30 minutes every day during 8 weeks
  Interventions: Device: transvaginal placebo device

INTERVENTIONS:
Device: transvaginal placebo device — Use of a transvaginal placebo home use programmable device used 30 minutes every day during 8 weeks
  Arms: 2
Device: transvaginal electrical stimulation device — Use of a transvaginal electrical stimulation home use programmable device used 30 minutes every day during 8 weeks
  Arms: 1

SUMMARY:
To compare the effectiveness of a transvaginal electrical stimulation by a home use programmable device to a placebo device for urinary incontinence in women

ELIGIBILITY:
Inclusion Criteria:

* >=18 years old
* Signed informed consent form
* Women with urinary stress incontinence defined as follow
* Involuntary loss of urine during increased abdominal pressure. In case of mix urinary incontinence (i.e., stress urinary incontinence associated to urge urinary incontinence) the discomfort related to stress incontinence as evaluated on a 0 (no discomfort) to 100 (maximum discomfort) visual analogic scale is higher for stress incontinence than for urge incontinence symptoms.
* closure pressure between 10 and 60 cm H2O
* the discomfort related to stress incontinence as evaluated on a 0 (no discomfort) to 100 (maximum discomfort) visual analogical scale is higher than 40/100
* Patients never treated with transvaginal electrical stimulation
* Vaginal muscle strength less than 3/5 on the muscular testing
* Positive Pad test (>2 g of leakage measure by pad test with standardised bladder volume)

Exclusion Criteria:

* Patient refusing to sign the consent form
* patient unable to understand or follow the protocol
* inadequate cognitive ability
* patient participating in another research protocol within the 3 previous months
* pregnancy
* women with no contraception
* pacemaker
* history of recent (< 1 year) transvaginal electrical stimulation treatment at home
* urinary incontinence other than stress incontinence
* neurological disease
* permanent metrorrhagia
* ongoing urinary tract infections
* vaginal prolapse > 2
* untreated atrophic vaginitis
* history of surgical treatment for urinary stress incontinence or genital prolapse
* recent pelvic surgery (<6 months)
* anatomic defect that preclude the use of the device
* genitourinary cancer or colic cancer
* patient already treated for urinary stress incontinence
* Recent oestrogen treatment (less than 3 weeks)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Number of urinary stress incontinence episodes measured by patients on a 7 days diary at 8 weeks | 8 weeks
Assessment of the discomfort linked to urinary stress incontinence occurring the previous week assessed on a 0 - 100 visual analog scale at 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Urodynamic investigation | 4 and 8 weeks
Standardised Pad test | 4 and 8 weeks
Number of severe urinary stress incontinence episodes | 4 and 8 weeks
Number of sanitary napkins used | 4 and 8 weeks
Leakage index | 4 and 8 weeks
Subjective appreciation of patients | 4 and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre européen d'explorations gynécologiques, Paris, France